CLINICAL TRIAL: NCT02175186
Title: Protective Effect of ALBIS on Gastroduodenal Mucosal Injury in Patients Receiving Dual Antiplatelet Therapy After Percutaneous Coronary Intervention
Brief Title: Effect of ALBIS on Gastroduodenal Mucosal Injury in Patients Receiving Dual Antiplatelet Therapy After Percutaneous Coronary Intervention
Acronym: DAPTALBIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Young-Hak Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCCV 2014-05
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Gastritis; Gastroduodenal Ulcer
Keywords: Gastritis; Gastroduodenal Ulcer; Percutaneous Coronary Revascularization; Dual Antiplatelet Therapy
MeSH Terms: conditions — Gastritis; Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALBIS (Experimental): Albis Tab 2 tab twice a day 12weeks
  Interventions: Drug: ALBIS
- Placebo (Placebo Comparator): placebo Tab 2 tab twice a day 12weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALBIS
  Arms: ALBIS
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate effectiveness of ALBIS on Gastroduodenal Mucosal Injury in Patients Receiving Dual Antiplatelet Therapy after Percutaneous Coronary Intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years
* Patients undergoing percutaneous coronary intervention and need to take dual antiplatelet therapy continuously at least 12weeks
* Modified Lanza Score grade 0-1 measured by upper gastrointestinal endoscopy
* mild gastrointestinal symptom
* Creatinen in blood ≤ 3mg/dl
* BUN ≤ 50mg/dl
* Birilubin ≤ 3mg/dl
* AST and ALT ≤ 80U/L

Exclusion Criteria:

* Pregnant or breast feeding
* History of Stomach or esophagus surgery
* Peptic ulcer or reflux esophagitis
* Zollinger-Ellison syndrome or primary esophageal motility disorders
* Malignant tumor
* Bleeding tendency or coagulopathy
* Contraindication of ALBIS
* Long term use of aspirin or P2Y12 receptor antagonist within 1month
* Patients who tool medicine such as PPI, APA,H2blocker, Muscarine receptor antagonist, anti-gastic agent, antacid, anticaogulant, Bisphosphonate agents, Cytotoxic drug, NSAID, adrenal cortex hormone agents (topical treatment is allowed)
* Terminal patient

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of gastric ulcer | 12weeks
  defined as a mucosal break of at least 5 mm in diameter(measured by gastrointestinal endoscopy) with depth, at 12weeks

SECONDARY OUTCOMES:
Incidence of gastritis | 12weeks
  defined as Modified Lanza Score(MLS) grade 2~4(measured by gastrointestinal endoscopy)at 12weeks
The Endoscopic improvement rate of hemorrhage | 12weeks
  defined as Modified Lanza Score(MLS) grade
The Endoscopic improvement rate of subjective symptom | 12weeks
Total amount of antacid used during study period | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hak Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea